CLINICAL TRIAL: NCT03404700
Title: Determining Dietary Pattern Accompanying Egg Intake Using Remote Food Photography Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Pennington Biomedical Research Center (Other); American Egg Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB2017-215
Record Dates: First submitted 2017-12-22; First posted 2018-01-19 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Eggs, saturated fat, insulin resistance,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The proposed study will comprise of two parts: Part I: an observational study based on ecological momentary assessment, and Part II: a randomized partial crossover clinical trial. Same subjects will participate in both parts of the study.
  In the observational study, the dietary intake of the subjects will be evaluated using an ecological momentary assessment approach for 7 days. In the randomized partial crossover clinical trial, four test breakfasts will be administered so that each subject will get exposed to only two out of the four diets (thus, partial crossover). Therefore, there will be six possible combinations of diets (i.e. 4! / 2! [4-2]!) and 12 possible ordered combinations (i.e. permutations; 4! / [4-2]!) of diets. Four subjects will be randomly assigned to each of these 12 possible ordered combinations of diets. Thus, the total sample size will be 48 (i.e. n = 4x12).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1:Test breakfast A and B (Experimental): *Please note: Part I of the study does not have separate groups. All subjects will undergo RFPM. The description of groups presented below is for part II of the study.
  Subjects will have egg breakfast(test breakfast A) and egg breakfast with high saturated fat (test breakfast B) in any order.
  Interventions: Behavioral: Egg breakfast; Behavioral: Egg breakfast with high saturated fat
- Group 2:Test breakfast A and C (Experimental): Subjects will have egg breakfast and (test breakfast A) and cereal breakfast (test breakfast C) in any order.
  Interventions: Behavioral: Egg breakfast; Behavioral: Cereal breakfast
- Group 3:Test breakfast A and D (Experimental): Subjects will have egg breakfast (test breakfast A) and cereal breakfast (test breakfast C) in any order.
  Interventions: Behavioral: Egg breakfast; Behavioral: Cereal breakfast with high saturated fat
- Group 4:Test breakfast B and C (Experimental): Subjects will have egg breakfast with high saturated fat (test breakfast B) and cereal breakfast (test breakfast C) in any order.
  Interventions: Behavioral: Egg breakfast with high saturated fat; Behavioral: Cereal breakfast
- Group 5:Test breakfast B and D (Experimental): Subjects will have egg breakfast with high saturated fat (test breakfast B) and cereal breakfast with high saturated fat (test breakfast D) in any order.
  Interventions: Behavioral: Egg breakfast with high saturated fat; Behavioral: Cereal breakfast with high saturated fat
- Group 6:Test breakfast C and D (Experimental): Subjects will have cereal breakfast (test breakfast C) and cereal breakfast with high saturated fat (test breakfast D) in any order
  Interventions: Behavioral: Cereal breakfast; Behavioral: Cereal breakfast with high saturated fat

INTERVENTIONS:
Behavioral: Egg breakfast — Containing:2 Scrambled Eggs, 120 mL Skim Milk, 2 Slices Nature's Own Double Fiber Wheat Bread, 30g Margarine, 18g Smuckers Strawberry Jam
  10 g of Margarine, 18 g of Smuckers® Strawberry Jam
  Other Names: Breakfast A
  Arms: Group 1:Test breakfast A and B; Group 2:Test breakfast A and C; Group 3:Test breakfast A and D
Behavioral: Egg breakfast with high saturated fat — Containing:2 Scrambled Eggs, 120 mL 2% milk, 2 Slices Nature's Own Double Fiber Wheat Bread, 15 g Butter, 15g Smuckers Strawberry Jam
  Other Names: Breakfast B
  Arms: Group 1:Test breakfast A and B; Group 4:Test breakfast B and C; Group 5:Test breakfast B and D
Behavioral: Cereal breakfast — Containing: 1c Special K ready-to-eat (RTE) High Protein Cereal, 200 mL Silk Original Soy milk, 1 Slice Mrs. Bairds Extra Thin Bread, 35g Margarine, 10 g Smuckers Sugar Free Strawberry Jam
  Other Names: Breakfast C
  Arms: Group 2:Test breakfast A and C; Group 4:Test breakfast B and C; Group 6:Test breakfast C and D
Behavioral: Cereal breakfast with high saturated fat — Containing: 1c Special K ready-to-eat (RTE) High Protein Cereal, 200 mL Silk Original Soy milk, 1/2 Slice Arnold Double Protein Whole Grain Bread, 15 g Butter
  Other Names: Breakfast D
  Arms: Group 3:Test breakfast A and D; Group 5:Test breakfast B and D; Group 6:Test breakfast C and D

SUMMARY:
Recent epidemiological studies show that egg consumption is associated with insulin resistance and altered glycemic control. For this study, the investigators hypothesize that this association is due to dietary patterns associated with egg consumption, such as saturated fat, and not the consumption of eggs per se. This study will be conducted in two parts that will be conducted simultaneously. Part I will utilize an ecological momentary assessment approach in which dietary patterns associated with egg intake will be determined using an objective measurement of food intake called remote food photography method. In Part II, a randomized partial crossover study will be conducted on the same sample of subjects to test the effects of egg consumption, saturated fat consumption, and consumption of the combination of eggs and saturated fat on glucose, insulin, and hunger and satiety hormone levels.

DETAILED DESCRIPTION:
Eggs are nutrient dense, convenient, affordable, and provide key macro and micronutrients in one's diet. Despite having a lot of benefits of consuming eggs in relation to health recent epidemiological studies raise health concerns about egg intake for subgroups of people. For instance, under free-living conditions, higher egg intake is associated with increased cardiovascular disease (CVD) risk in diabetic individuals as well as increased risk of developing type 2 diabetes. However, these studies do not establish that egg consumption "causes" health issues.

It is also possible that the association of egg intake with increased CVD risk in diabetics, or with a greater risk of developing diabetes, is simply due to the other foods that people usually eat with eggs, such as saturated fats, and not due to eggs per se.

For part I, the investigators propose to test this hypothesis by determining the food intake of 48 non-diabetic individuals under free-living conditions using the remote food photography method (RFPM), which uses smartphone technology. The frequency of egg consumption will be obtained using a food frequency questionnaire (FFQ). In addition, participants will record their food intake using food record diary and a 24-hour food recall method. Energy intake information gathered from RFPM will be compared with the 7-day food record and the 24-hour recall.

Next, for part II, the same study participants will be offered four separate test breakfasts of similar calories, containing 1) Eggs; 2) Eggs with a high amount of saturated fat; 3) Cereal breakfast (neither eggs nor saturated fat); or 4) Cereal breakfast with a high amount of saturated fat. Alteration of blood glucose, insulin, hunger, and satiety hormones (ghrelin, PYY, GLP-1), and metabolic rate will be measured before and after each breakfast in part II.

The investigators expect to determine if the purported association of eggs to alterations in glucose control and related metabolic alterations are independent of eggs, but mainly due to saturated fat is eaten along with eggs rather than the egg consumption itself.

ELIGIBILITY:
Inclusion Criteria:

* 48 non-diabetic individuals (fasting glucose < 126 mg/dL)
* Male or female
* BMI from greater or equal to 20 to lesser or equal 60 kg/m2
* Age: 18 - 65 years

Exclusion Criteria:

* Diabetes
* On antidiabetes medication
* Pregnant or lactating females
* Having a history of gestational diabetes
* Having an unstable cardiac condition
* Having a major systemic illness
* Having a history of drug abuse
* Having a history of eating disorders
* Having uncontrolled hypothyroidism
* Having familial hyperlipidemias
* Having allergies sensitivity to or dislike of eggs
* Consumption of < 1 egg per week
* Attempting to lose weight
* On medications that may influence or inhibit appetite, sensory functioning, or hormone signaling- e.g. antibiotics, anti-depressants, obesity medications. Weight loss > 5% in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Difference of energy intake (kcal) in meals containing eggs as compared to meals that do not contain eggs | Day 1-7 of the ecological momentary assessment part (Part I) of the study
  Energy intake will be determined using Remote Food Photography Method (RFPM) and the meals of all test subjects will be categorized based on the presence or the absence of eggs in the meals.
Difference of energy intake (kcal) in high egg consumers as compared to low egg consumers | Day 1-7 of the ecological momentary assessment part (Part I) of the study
  Comparison of mean daily energy intake as measured by Remote Food Photography Method (RFPM) between high egg consumers and low egg consumers identified by providing a food frequency questionnaire (FFQ).
Difference of saturated fat (g) intake in meals containing eggs as compared to meals that do not contain eggs | Day 1-7 of the ecological momentary assessment part (Part I) of the study
  Saturated fat intake will be determined using Remote Food Photography Method (RFPM) and the meals of all test subjects will be categorized based on the presence or the absence of eggs in the meals.
Difference of saturated fat (g) intake in high egg consumers as compared to low egg consumers | Day 1-7 of the ecological momentary assessment part (Part I) of the study
  Comparison of saturated fat intake as measured by Remote Food Photography Method (RFPM) between high egg consumers and low egg consumers identified by providing a food frequency questionnaire (FFQ).
Difference of blood glucose levels compared between different test breakfasts | Changes in concentration (area under the curve; AUC) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts.
Difference of insulin levels compared between different test breakfasts | Changes in concentration (area under the curve; AUC) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts.

SECONDARY OUTCOMES:
Difference of subjective hunger level compared between different test breakfasts | Changes in scores (arbitrary units AU) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts.
Difference of subjective satiety level compared between different test breakfasts | Changes in scores (arbitrary units AU) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts.
Difference of objective hunger compared between different test breakfasts | Changes in concentration (area under the curve AUC) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts by measuring serum ghrelin levels.
Difference of objective satiety compared between different test breakfasts using serum Glucagon-like peptide-1 (GLP-1) levels | Changes in concentration (area under the curve AUC) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts by measuring serum GLP-1 levels.
Difference of objective satiety compared between different test breakfasts using serum Peptide YY (PYY 3-36) levels | Changes in concentration (area under the curve AUC) from 30 minutes prior to breakfast to 180 minutes after consumption of test breakfasts (Part II of the study)
  This will be measured on visit 1 and 2 after providing test breakfasts by measuring serum PYY 3-36 levels.
Difference of HbA1c levels in high egg consumers as compared to low egg consumers | Changes in blood concentration (arbitrary units AU) on visit 1 (Part II of the study)
  This will be measured by taking blood on the visit 1.
Difference in Homeostasis Model Assessment-Insulin resistance (HOMA-IR) compared between different test breakfasts | Changes in HOMA-IR values (arbitrary units AU) on visit 1 and 2 after providing test breakfasts (Part II of the study)
  This will be calculated using blood glucose and insulin levels.
Difference in Resting Metabolic Rate (RMR) compared between different test breakfasts | Changes in RMR (kcal/24hrs) on visit 1 and 2 following each test breakfast ( Part II of the study)
  RMR will be assessed following different test breakfasts on visit 1 and 2.
Difference in total energy intake (kcal) compared between Remote Food Photography Method (RFPM), 7-day food record and 24-hour recall | Day 1-7 of the ecological momentary assessment part (Part I) of the study
  Comparison of mean energy intake as determined by RFPM with mean energy intake determined by 7-day food record and a single 24-hour recall.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu FB, Stampfer MJ, Rimm EB, Manson JE, Ascherio A, Colditz GA, Rosner BA, Spiegelman D, Speizer FE, Sacks FM, Hennekens CH, Willett WC. A prospective study of egg consumption and risk of cardiovascular disease in men and women. JAMA. 1999 Apr 21;281(15):1387-94. doi: 10.1001/jama.281.15.1387. PMID 10217054
- [Background] Shin JY, Xun P, Nakamura Y, He K. Egg consumption in relation to risk of cardiovascular disease and diabetes: a systematic review and meta-analysis. Am J Clin Nutr. 2013 Jul;98(1):146-59. doi: 10.3945/ajcn.112.051318. Epub 2013 May 15. PMID 23676423
- [Background] Djousse L, Gaziano JM, Buring JE, Lee IM. Egg consumption and risk of type 2 diabetes in men and women. Diabetes Care. 2009 Feb;32(2):295-300. doi: 10.2337/dc08-1271. Epub 2008 Nov 18. PMID 19017774
- [Background] Wallin A, Forouhi NG, Wolk A, Larsson SC. Egg consumption and risk of type 2 diabetes: a prospective study and dose-response meta-analysis. Diabetologia. 2016 Jun;59(6):1204-13. doi: 10.1007/s00125-016-3923-6. Epub 2016 Mar 18. PMID 26993632
- [Background] Martin CK, Correa JB, Han H, Allen HR, Rood JC, Champagne CM, Gunturk BK, Bray GA. Validity of the Remote Food Photography Method (RFPM) for estimating energy and nutrient intake in near real-time. Obesity (Silver Spring). 2012 Apr;20(4):891-9. doi: 10.1038/oby.2011.344. Epub 2011 Dec 1. PMID 22134199
- [Derived] Dhanasekara CS, Dawson JA, Martin CK, Dhurandhar NV. No association between consumption of eggs with energy or macronutrient intake: Objective evidence from the remote food photography method. Diabetes Metab Syndr. 2021 Jan-Feb;15(1):313-318. doi: 10.1016/j.dsx.2021.01.010. Epub 2021 Jan 15. PMID 33486223

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03404700/Prot_SAP_ICF_002.pdf